CLINICAL TRIAL: NCT04696627
Title: Long-term Complications of Unintentional Dural Puncture During Labour Epidurals and Epidural Blood Patch.
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20-03
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-02

CONDITIONS: Post-Dural Puncture Headache; Chronic Headache
Keywords: post-dural puncture headache; labour epidural; chronic headache; chronic backache
MeSH Terms: conditions — Post-Dural Puncture Headache; Headache Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dural puncture: Patients with well-documented recognized unintentional dural punctures during their labor epidural insertion at Mount Sinai Hospital from January 2015 to December 2019.
  Interventions: Other: Questionnaire
- Dural puncture with blood patch: Patients with well-documented recognized unintentional dural punctures during their labor epidural insertion at Mount Sinai Hospital from January 2015 to December 2019 that were treated with an epidural blood patch.
  Interventions: Other: Questionnaire
- No dural puncture: Patients who did not have recognized unintentional dural punctures during their labor epidural insertion at Mount Sinai Hospital from January 2015 to December 2019.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Participants from all 3 groups will be interviewed

SUMMARY:
The investigators plan to evaluate long-term consequences of unintentional dural puncture in women who had this complication during labor epidural insertion at Mount Sinai Hospital. A dural puncture is the perforation of the dura mater (one of the layers protecting the brain and the spinal cord) by the needle that is used to find and place a catheter in the epidural space. A puncture will cause a leakage of cerebrospinal fluid through the dura that results in an acute and usually self-limited headache in half of patients who have this complication. The usual treatment for this complication is conservative with the use of oral medications like acetaminophen, anti-inflammatory and narcotics. In the severely symptomatic patient, the injection of blood in the epidural space is a more invasive approach performed to "patch" the hole that was created in the dura (epidural blood patch). The objective is to determine whether or not there is a risk of developing long-term effects from the unintentional dural puncture and its treatment by epidural blood patch by comparing women who had a dural puncture during their labour epidural insertion with or without an epidural blood patch with women who received an epidural but did not have a dural puncture during the same period of time.

The hypothesis is that women who had unintentional dural punctures during epidural insertion will develop long-term effects such as chronic headache, chronic backache, chronic auditory or visual disturbances and chronic disability more frequently than women who received an epidural but did not sustain a dural puncture. The investigators also hypothesize that the use of epidural blood patch may change the course of these complications.

DETAILED DESCRIPTION:
The investigators will study women who have sustained an unintentional dural puncture at least one year prior to the start date of the study, and the investigators will study cases occurring during a period of 5 years. These women will be matched by type of procedure (labor epidural), month of delivery and age with women who have received an epidural but did not sustain an unintentional dural puncture. The group of women who sustained dural punctures will be further divided into two groups, whether they have received epidural blood patch or not, to study the influence of the epidural blood patch on the outcomes. Women will have their anesthetic records reviewed to collect data on the anesthetic technique, presence of a dural puncture and treatment if applicable. All patients who qualify will be contacted and invited to take part in this study. Those consenting to the study will be interviewed by phone or answer the survey electronically. During the interview, they will answer questions derived from validated questionnaires for the majority of our outcomes of interest. In the few outcomes where a validated questionnaire does not exist, the investigators will search for our endpoint with dichotomic (yes/no) questions. The investigators will then compare the data gathered in the three different groups to validate or invalidate our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* All patients with well-documented recognized unintentional dural punctures during their labor epidural insertion at Mount Sinai Hospital from January 2015 to December 2019 will be approached for enrollment. Control patients who received labor epidural matched by month of delivery and age will also be approached for enrollment.

Exclusion Criteria:

* Patients with preexisting symptoms of chronic headache, or any of the secondary outcomes prior to the unintentional dural puncture will be excluded from this study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with labour epidurals inserted at Mount Sinai hospital from January 2015 to December 2019 with well-documented recognized unintentional dural punctures will be invited to participate.
  Control patients who received labor epidural matched by month of delivery, age, and body mass index (grouped as either below or above a body mass index of 40) will also be approached for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Presence of Chronic headache - questionnaire | 3 months
  The presence of chronic headache defined as pain that lasts or recurs for more than three months.

SECONDARY OUTCOMES:
Presence of Chronic lower back pain - questionnaire | 3 months
  Presence of Chronic lower back pain, with or without neuropathic features, defined as pain that lasts or recurs for more than three months.
Presence of Chronic auditory impairment - questionnaire | 3 months
  The presence of auditory impairment defined as impairment that lasts or recurs for more than three months.
Presence of Chronic visual impairment - questionnaire | 3 months
  The presence of chronic visual impairment defined as impairment that lasts or recurs for more than three months.
Medical interventions for pain/impairment - questionnaire | 3 months
  The treatment of any pain/impairment described by the patient.
Pain disability index - questionnaire | 3 months
  Whether any pain/impairment described by the patient affects activities of daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada